CLINICAL TRIAL: NCT04770974
Title: Definition of Tumor Bio-markers and Physical-spectroscopic Differences Between Healthy Urothelial Tissue Healthy and Urothelial Cancer
Brief Title: Urothelial Cancer Tumor Bio-markers and Physical-spectroscopic Characteristic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Florence (Other)
Collaborators: University of Milano Bicocca (Other); Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government); Careggi Hospital (Other)
Responsible Party: Principal Investigator, Simone Morselli, PhD Student, University of Florence
Other Study IDs: 17852_bio
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Urothelial Carcinoma; Bladder Cancer; Urothelial Neoplasm; Urothelial Carcinoma Bladder; Urothelial Carcinoma in Situ
Keywords: spectroscopy; bladder cancer; urothelial carcinoma; tumor biomarkers; metabolomic; proteomic
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Urothelial Carcinoma: Patients over the age of 18 known for urological interventions for the following pathologies will be considered for enrollment in the group of cases:
  - Bladder cancer
  The exclusion criteria will be:
  * Age under 18
  * Pregnancy
  * Lack of informed consent
  * Inability to provide informed consent
  Patients included in the study, who meet the inclusion criteria, have an operative note for:
  * Transurethral Resection of Bladder Neoplasia (TURBT)
  * Radical Cystectomy for Bladder Neoplasia
  Interventions: Other: Biomarkers and proteomics

INTERVENTIONS:
Other: Biomarkers and proteomics — Biomolecular, proteomic, metabolomic and spectroscopy characterization of urothelial bladder neoplasia, on a 3D culture model (organoid) obtained from bladder tumor tissue

SUMMARY:
Our multicenter observational study is a non-profit prospective study. The study was born from the Amplitude Project, which comprise the SOD of Minimally Invasive Robotic Urological Surgery and Renal Transplants of AOU Careggi with the University of Florence, as well as with the National Research Council (CNR) and the University of Milan Bicocca (UNIMIB) The study consists of a phase of enrollment of patients who will be admitted to the SOD of Mini Invasive Robotic Urological Surgery and Renal Transplantation of AOU Careggi. Enrollment in the study does not alter normal clinical practice and does not involve additional risks for patients. Patients will have to meet the inclusion and exclusion criteria of the study and will be enrolled sequentially, until the established sample size is reached. Patients undergoing surgery for the removal of bladder neoplasm, be it endoscopic or surgical with radical intent (cystectomy), will be taken a fragment of tumor bladder tissue, on which histopathological analysis will be performed. In patients undergoing radical cystectomy only, a fragment of healthy urothelial tissue, free from neoplasia, will also be removed. The samples will be performed in patients under general and / or spinal anesthesia in case of TURB, thus not causing pain or discomfort to the patient, or ex-vivo on the operative piece in case of radical cystectomy, without causing further damage or pain to the patient. From these samples, specially stored in solutions that keep their characteristics unaltered, a 3D culture model (organoid) will be obtained both from cells obtained from bladder cancer and from healthy tissue on which biomolecular, metabolomic and spectroscopic characterization studies will be tested and carried out. with a view to staging and grading bladder neoplasia.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Bladder Cancer diagnosis
* Capability to express informed consent

Exclusion Criteria:

* Age under 18
* Pregnancy
* Lack of informed consent
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo a surgical intervention for bladder cancer will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-12-10 (Actual); Primary Completion 2022-12-07 (Estimated); Study Completion 2022-12-07 (Estimated)

PRIMARY OUTCOMES:
Metabolomic | Enrollment
  Metabolomic characteristic of bladder cancer
Spectroscopy | Enrollment
  Spectroscopical characteristic of bladder cancer

SECONDARY OUTCOMES:
Progression | Seven years
  Comparison between different progression pattern among bladder cancer
Response to treatments | Seven years
  Comparison between different treatment response pattern among bladder cancer
Survival | Seven years
  Comparison between different survival outcomes among bladder cancer
Transcriptomic | Enrollment
  Transcriptomic characteristic of bladder cancer

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Serni, Prof, Principal Investigator — University of Florence; Mauro Gacci, MD, Principal Investigator — AOU Careggi
Locations (1):
- Careggi Hospital, Florence, Tuscany, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baria E, Morselli S, Anand S, Fantechi R, Nesi G, Gacci M, Carini M, Serni S, Cicchi R, Pavone FS. Label-free grading and staging of urothelial carcinoma through multimodal fibre-probe spectroscopy. J Biophotonics. 2019 Nov;12(11):e201900087. doi: 10.1002/jbio.201900087. Epub 2019 Aug 13. PMID 31343832
- See also: Related Info — https://www.amplitude-imaging.com/